CLINICAL TRIAL: NCT05120986
Title: Sensor: ENhancing aSthma carE - An Observational Prospective Study to Characterize Patients Initiating Indacaterol + Glycopyrronium Bromide + Mometasone Furoate (Enerzair® Breezhaler®), With or Without Sensor, as a Maintenance Treatment for Asthma
Brief Title: An Observational Prospective Study to Characterize Patients Initiating Enerzair® Breezhaler®, With or Without Sensor, as a Maintenance Treatment for Asthma
Acronym: SENSE
Status: Withdrawn | Type: Observational
Why Stopped: Novartis Farma - Produtos Farmaceuticos S.A. no longer commercializes the product.
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Other Study IDs: CQVM149BPT01
Record Dates: First submitted 2021-11-03; First posted 2021-11-16 (Actual); Last update posted 2022-04-04 (Actual); Status verified 2022-03

CONDITIONS: Asthma
Keywords: Asthma; SENSE study; Enerzair; Breezhaler; maintenance treatment
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (2):
- IND/GLY/MF with sensor: Patients prescribed with indacaterol acetate, glycopyrronium bromide and mometasone furoate with sensor
  Interventions: Other: IND/GLY/MF
- IND/GLY/MF without sensor: Patients prescribed with indacaterol acetate, glycopyrronium bromide and mometasone furoate without sensor
  Interventions: Other: IND/GLY/MF

INTERVENTIONS:
Other: IND/GLY/MF — Prospective observational cohort study. There is no treatment allocation. Patients will be invited to participate in the study when attending participating community pharmacies with a first prescription of IND/GLY/MF with sensor or IND/GLY/MF without sensor
  Other Names: Enerzair® Breezhaler®

SUMMARY:
This is an observational, descriptive, open-label, prospective, 6-month study including a group of patients with a first prescription of IND/GLY/MF with sensor and a group with a first prescription of IND/GLY/MF without sensor.

DETAILED DESCRIPTION:
Patients will be invited prospectively and sequentially to participate in the study when attending a participating community pharmacy with a first prescription of IND/GLY/MF with sensor or IND/GLY/MF without sensor. Therefore, the invitation for the patient to participate in the study will occur only after the therapeutic decision has taken place

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients aged ≥18 years
* Self-reported diagnosis of asthma
* Individual filling a first prescription of IND/GLY/MF with or without sensor in a participating community pharmacy for himself/herself (excluding caregivers).
* Individual capable and willing to perform the study assessments.

Exclusion Criteria:

* No exclusion criteria.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with a first prescription of IND/GLY/MF with sensor and a group of patients with a first prescription of IND/GLY/MF without sensor at a community pharmacy setting.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2022-02-15 (Estimated); Primary Completion 2023-05-15 (Estimated); Study Completion 2023-05-15 (Estimated)

PRIMARY OUTCOMES:
Baseline sociodemographic - living status | Baseline
  Assess if the patient lives alone:
  * Yes
  * No
  * Don't know/ Don't answer
Baseline sociodemographic - household income | Baseline
  Patient's household net income level:
  * <665 €
  * [665€ to 1000€[
  * [1000€ to 1200€[
  * [1400€ to 1700€[
  * [1700€ to 2000€[
  * [2000€ to 2700€[
  * ≥2700€
  * Don't know/Don't answer
Baseline sociodemographic - educational level | Baseline
  Patient's highest completed educational level:
  * None
  * I - Basic education (4 years)
  * II - Basic education (6 years)
  * III - Basic education (9 years)
  * Upper secondary education or equivalent (12 years)
  * Bachelor/ University Degree
  * Don't know/Don't answer
Baseline sociodemographic - employment status | Baseline
  Patient Employment status:
  * Employed. Number of hours per week.
  * Unemployed
  * Student
  * Retired
  * Other. Specify.
  * Don't know/Don't answer
clinical characteristics - body mass index | Baseline
  body mass index will be provided
clinical characteristics - smoking status | Baseline
  Patient smoking status:
  * Never smoked
  * Ex-smoker
  * Smoker
  * Don't know/Don't answer
clinical characteristics - comorbidities | Baseline
  Patient comorbidities:
  * Allergic rhinitis
  * Rhinosinusitis
  * Allergic conjunctivitis
  * Sleep disorders
  * Anxiety
  * Depression
  * Other. Specify
clinical characteristics - duration of disease | Baseline
  duration of disease will be provided
clinical characteristics - age at asthma diagnosis | Baseline
  Age when asthma was diagnosed:
  * Years
  * Unknown/cannot remember
clinical characteristics - asthma-related hospitalizations | Baseline
  Number of hospitalizations:
  * n of hospitalizations
  * Don't know/Don't answer
clinical characteristics - emergency admissions and non-scheduled visits in the previous 12 months | Baseline
  Number of appointments:
  * number of scheduled asthma physician's appointments
  * number of unscheduled asthma physician's appointments
  * Don't know/Don't answer
clinical characteristics - ACT score | Baseline
  The Asthma Control Test (ACT) contains 5 questions that are related to the frequency of both asthma symptoms and required rescue medication use during the previous 4 weeks. The scores in the ACT range from 5 (worse control) to 25 (total control)
clinical characteristics - TAI score | Baseline
  The TAI questionnaire was developed to measure self-reported adherence to inhaler devices and help clinicians to evaluate non-adherence barriers related to inhaled therapy in adult patients with asthma or chronic obstructive pulmonary disease.
  The interpretation of adherence based on the 10-item TAI, scoring is that an overall score of 50 points highlights good adherence, while a score of between 46 to 49 points denotes intermediate adherence. A total score ≤ 45 points indicates poor adherence
clinical characteristics - last asthma treatment | Baseline
  International Nonproprietary Name (INN) of Last asthma medication

SECONDARY OUTCOMES:
Changes from baseline in self-reported adherence - TAI questionnaire score | Baseline, month 3, month 6
  The TAI questionnaire was developed to measure self-reported adherence to inhaler devices and help clinicians to evaluate non-adherence barriers related to inhaled therapy in adult patients with asthma or chronic obstructive pulmonary disease.
  The interpretation of adherence based on the 10-item TAI, scoring is that an overall score of 50 points highlights good adherence, while a score of between 46 to 49 points denotes intermediate adherence. A total score ≤ 45 points indicates poor adherence
Changes from baseline in self-reported adherence - asthma control test (ACT) score | Baseline, month 3, month 6
  The Asthma Control Test (ACT) contains 5 questions that are related to the frequency of both asthma symptoms and required rescue medication use during the previous 4 weeks. The scores in the ACT range from 5 (worse control) to 25 (total control)
Adherence from the app (percentage) | Month 3, month 6
  Adherence over last month to be measured using a scale from 0 to 100
Asthma control from the app (category) | Month 3, month 6
  Asthma control over last month:
  * Well controlled
  * Not properly controlled
  * Poorly controlled
  * Unknown
Rescue medication from the app | Month 3, Month 6
  Rescue medication over last month (n days):
  * N days
  * N days over the night period
Percentage of patients in treatment | month 3, month 6
  Percentage of patients in treatment will be provided
Reasons for discontinuation and treatment switch | month 3, month 6
  Reason for treatment discontinuation:
  * Tolerability
  * Loss of efficacy
  * Price
  * Problems with medication use
  * Following emergency/ hospitalization
  * Condition improved
  * Other. Specify.
  * Don't know/Don't answer
Change from baseline in number of hospitalizations | Baseline, month 3, month 6
  Number of hospitalizations and nights:
  * n of hospitalizations
  * n of nights
  * Don't know/Don't answer
Change from baseline in number of emergency room visits | Baseline, month 3, month 6
  Number of emergency room visits:
  * n (visits)
  * Don't know/don't answer
Change from baseline in number of scheduled and non-scheduled medical visits | Baseline, month 3, month 6
  Number of appointments:
  * n of scheduled appointments
  * n of unscheduled appointments
  * Don't know/ Don't answer
Change from baseline in number of work hours/days missed | Baseline, month 3, month 5
  How many hours/days the patient missed work or was delayed:
  * n (days)
  * Not applicable
Percentage of patients by level of treatment satisfaction | month 3, month 6
  Treatment satisfaction:
  Very satisfied
  * Satisfied
  * Not Satisfied/unsatisfied
  * Unsatisfied
  * Very Unsatisfied
Percentage of patients who downloaded the app in the group of IND/GLY/MF with sensor. | month 3, month 6
  Patient downloaded the app:
  * Yes
  * No
percentage of patients with a valid app report in the group of IND/GLY/MF with sensor. | month 3, month 6
  Number of patients that downloaded the app
percentage of patients reporting ease to use and understand how to use the sensor and the app in the group of IND/GLY/MF with sensor | month 3, month 6
  Ease to use the app/sensor:
  * Yes
  * No
  * Don't know/Don't answer
percentage of patients reporting usefulness of the sensor/app reports in asthma control and treatmen in the group of IND/GLY/MF with sensor.t | month 3, month 6
  Usefulness of the app report in learning about their asthma:
  * Yes
  * No
  * Don't know/Don't answer
Percentage of patients with desire to continue using sensor/app in the group of IND/GLY/MF with sensor. | month 3, month 6
  Desire to continue using the app:
  * Yes
  * No
  * Don't know/Don't answer
Percentage of patients with fair acquisition value for sensor/app in the group of IND/GLY/MF with sensor | month 3, month 6
  Fair acquisition value of sensor/app:
  * 0 €
  * 1 to 5 €
  * 6 to 10€
  * 11 to 15 €
  * 16 to 20 €
  * More than 20 €

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmceuticals, Study Director — Novartis Pharmaceuticals

IPD SHARING:
Plan to Share IPD: No